CLINICAL TRIAL: NCT02453152
Title: Respiratory Muscle Function in Untreated X-Linked Myotubular Myopathy (XLMTM)
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: Audentes Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: IRB201500379
Record Dates: First submitted 2015-05-18; First posted 2015-05-25 (Estimated); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: X-linked Myotubular Myopathy
Keywords: myotubular myopathy; respiratory muscles; natural history
MeSH Terms: conditions — Myopathies, Structural, Congenital | interventions — Health Records, Personal; Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Males with X-linked myotubular myopathy: History and physical, Tidal breathing, Maximal respiratory pressures, Peak cough flow, Pediatric Evaluation of Disability Inventory, PedsQL Multidimensional Fatigue Scale, Review of ventilation requirements
  Interventions: Other: History and physical; Other: Tidal breathing; Other: Maximal respiratory pressures; Other: Peak cough flow; Other: Pediatric Evaluation of Disability Inventory; Other: PedsQL Multidimensional Fatigue Scale; Other: Review of ventilation requirements

INTERVENTIONS:
Other: History and physical — Subjects will undergo a physical exam and medical history review, including review of genetic test results.
Other: Tidal breathing — Subjects' breathing patterns will be evaluated at rest and at reduced/eliminated ventilator support.
Other: Maximal respiratory pressures — Subjects' strongest inspiratory and expiratory pressures will be measured.
  Other Names: MIP, MEP
Other: Peak cough flow — Subjects' strongest coughs will be measured.
Other: Pediatric Evaluation of Disability Inventory — Assesses the functional capabilities of children with disabilities.
  Other Names: PEDI
Other: PedsQL Multidimensional Fatigue Scale — Assesses general fatigue, sleep/rest fatigue, and cognitive fatigue.
Other: Review of ventilation requirements — Subjects's use of mechanical ventilation reviewed by the study team.

SUMMARY:
This study is a longitudinal study evaluating the severity and progression of respiratory muscle function in patients with X-Linked Myotubular Myopathy (XLMTM) aged 0-14.

DETAILED DESCRIPTION:
Subjects aged 0-7 will be evaluated every six months for a total of three evaluations (Baseline, Six-Month Visit, Twelve-Month Visit). Subjects aged 8-14 will be evaluated every twelve months for a total of two evaluations (Baseline, Twelve-Month Visit). Evaluations include medical history, physical exam, respiratory muscle tests, a qualitative interview related to the child's function and use of respiratory aids, and quality of life assessments.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have centronuclear myopathy resulting from an MTM1 genetic mutation.
* Patients who are between 0 and 14 years of age.

Exclusion Criteria:

* Patients without a confirmed genetic mutation.
* Patients unable to travel to the site for the study.
* Patients participating in an interventional treatment study for XLMTM at the time of enrollment.
* Patients who are unable to complete study procedures.
* Patients who have a condition that, in the opinion of the investigator, would make participation in this study unsafe.

Max Age: 14 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Study Population: Males with geneticially confirmed XLMTM
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2015-10; Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Change in baseline visit off-ventilator tolerance at 6 month visit and 12 month visit. | Change in baseline visit, at 6 month visit and 12 month visit

SECONDARY OUTCOMES:
Change in baseline visit maximal respiratory pressures at 6 month visit, and 12 month visit. | Change in baseline visit, at 6 month visit and 12 month visit
  Subject's maximal inspiratory and expiratory pressures.
Change in baseline peak cough flow at 6 month visit and 12 month visit. | Change in baseline visit, at 6 month visit and 12 month visit
  Subjects will be assessed on the ability to generate a cough and the strength of that cough.
Change in baseline tidal breathing at 6 month visit and 12 month visit. | Change in baseline visit, at 6 month visit and 12 month visit
  Subject's resting breathing pattern will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara K Smith, PT, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States